CLINICAL TRIAL: NCT05589051
Title: Effect of Alpha Hope Dietary Supplement on Biochemical Markers of Health and Computerized Tests of Cognitive Performance
Brief Title: Effect of Alpha Hope Dietary Supplement on Health and Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Calerie LLC (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of the College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO-FY2022-130
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Cognitive Change
Keywords: Alpha Hope; Pyrroloquinoline Quinone; Molecular Hydrogen

STUDY DESIGN:
Intervention Model Description: Subjects take randomly assigned condition for 4 weeks, then washout for 3 weeks before crossing over to other condition for 4 weeks.
Who Masked: Participant, Investigator
Masking Description: Tablets will be of similar appearance and provided in bottles labeled A and B
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpha Hope (Experimental): Each tablet contains 10 mg PQQ and 40 mg (19% DV) magnesium as well as malic acid, dextrose, adipic acid, citric acid, natural flavor, and blackberry leaf extract
  Interventions: Dietary Supplement: Drink
- Placebo (Placebo Comparator): Same formulation as experimental with 250 mg calcium carbonate replacing the magnesium and PQQ.
  Interventions: Dietary Supplement: Drink

INTERVENTIONS:
Dietary Supplement: Drink — Consume one tablet fully dissolved in 8 ounces. Take 2 tablets per day for adults (morning and evening) for 4 weeks

SUMMARY:
The purpose of the present research study is to evaluate the claims about the supplement influencing cognitive function that may impact performance on cognitive task and related biochemical measures. The synergistic administration of Pyrroloquinoline Quinone and molecular Hydrogen (in the form of Alpha Hope) will be evaluated in adults without a diagnosis of disease (i.e., otherwise healthy adults-the population the supplement is marketed to) on certain biochemical markers, subject's self-assessed wellness, and functional measurements determined via computer tests.

DETAILED DESCRIPTION:
Alpha Hope is a dietary supplement that contains Pyrroloquinoline Quinone and Magnesium-which has been shown to generate molecular hydrogen when mixed into water. Both Pyrroloquinoline Quinone and molecular hydrogen have been shown to exhibit antioxidant and anti-inflammatory capacities. Both Pyrroloquinoline Quinone and magnesium are widely used as dietary supplements, alone and in combination with other ingredients; however, to our knowledge, this is the first time that these two ingredients have been coupled together within one dietary supplement.

Previous research has demonstrated a wide range of health benefits from Pyrroloquinoline Quinone. Of particular interest, Pyrroloquinoline Quinone has been shown to improve cognition when supplemented at daily dosages similar to that proposed in the present study.

Molecular hydrogen has inherent anti-apoptosis, anti-inflammatory, and anti-oxidation properties and has therefore been studied in numerous animal studies, as well as human studies as a possible treatment for degenerative brain function. One method for generating molecular hydrogen, is using elemental magnesium, which reacts with water to generate molecular hydrogen.

The purpose of the present research study is to evaluate the claims about the supplement influencing cognitive function that may impact performance on cognitive task and related biochemical measures. The synergistic administration of Pyrroloquinoline Quinone and molecular Hydrogen (in the form of Alpha Hope) will be evaluated in adults without a diagnosis of disease -(i.e., otherwise healthy adults- the population the supplement is marketed to) on certain biochemical markers, subject's self-assessed wellness, and functional measurements determined via computer tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (no diagnosed disease, including but not limited to metabolic, cardiovascular disease, or neurological disease)
* Able to consume calcium carbonate (the placebo)
* able to fast overnight (>10 hrs)

Exclusion Criteria:

* tobacco user
* currently taking a physician recommended medication/dietary supplement for cognition or brain health, including donepezil (Aricept®), rivastigmine tartrate (Exelon®), galantamine HBr (Reminyl®), and memantine (Namenda®), modafinil (Provigil®), Ginkgo biloba, ginseng B vitamins, Vitamin E, omega-3 fatty acids, Vitamins A & C, Vitamin D, phosphatidylserine, phosphatidylcholine, or supplements with brain, cogni, neuro, or similar in their names.
* taking an over-the-counter medication or dietary supplement that can effect cognition/brain health, including Ginkgo biloba, ginseng B vitamins, Vitamin E, omega-3 fatty acids, Vitamins A & C, Vitamin D, phosphatidylserine, phosphatidylcholine, or supplements with brain, focus, memory, cogni, or neuro in their names.
* diagnosed with any of these conditions (contraindicative for calcium carbonate): high calcium levels (hypercalcemia), stomach/intestinal blockage, kidney disease (such as kidney stones) (Cleveland Clinic)
* taking any medication that interacts with calcium carbonate including ammonium chloride, methenamine, antibiotics like ciprofloxacin or tetracycline, captopril, delavirdine, gabapentin, iron supplements, medicines for fungal infections like ketoconazole and itraconazole, medicines for seizures like ethotoin and phenytoin, mycophenolate, quinidine, rosuvastatin, sucralfate, thyroid medicine (Cleveland Clinic)
* consumption of alcohol-containing beverages within 24 hours of testing
* consumption of caffeine within 24 hours of testing
* strenuous exercise within 24 hours of testing
* self-reported active infection or illness of any kind
* pregnant or lactating
* allergic or hypersensitive to any of the components of the supplement and placebo: PQQ, magnesium, malic acid, dextrose, adipic acid, citric acid, natural flavor, blackberry leaf extract, calcium carbonate

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Digit Symbol Substitution test | baseline
  Using the response key (at the top of the test), subjects select the corresponding number with a computer mouse that corresponds with the specific symbol displayed on the computer screen to obtain as many correct responses as they can within a set time frame (two minutes)
Digit Symbol Substitution test | 4 week timepoint
  Using the response key (at the top of the test), subjects select the corresponding number with a computer mouse that corresponds with the specific symbol displayed on the computer screen to obtain as many correct responses as they can within a set time frame (two minutes)
AX-Continuous Performance Test | baseline
  Subject press different keys on a keyboard to indicate if the stimulus is the target (AX) or non-target to measure accuracy and response time
AX-Continuous Performance Test | 4 week timepoint
  Subject press different keys on a keyboard to indicate if the stimulus is the target (AX) or non-target to measure accuracy and response time
Go/No-Go test | baseline
  Subjects press a key when Go is displayed and no key when No Go is displayed to test accuracy and reaction time.
Go/No-Go test | 4 week timepoint
  Subjects press a key when Go is displayed and no key when No Go is displayed to test accuracy and reaction time.
irisin | baseline
  Irisin is quantified from blood sample
irisin | 4 week timepoint
  Irisin is quantified from blood sample
brain-derived neurotrophic factor | baseline
  Brain-derived neurotrophic factor is quantified from blood sample
brain-derived neurotrophic factor | 4 week timepoint
  Brain-derived neurotrophic factor is quantified from blood sample
Fibroblast growth factor 21 | baseline
  Fibroblast growth factor 21 factor is quantified from blood sample
Fibroblast growth factor 21 | 4 week timepoint
  Fibroblast growth factor 21 factor is quantified from blood sample
Self-reported Wellness Assessment | baseline
  Subjects report their self-reported wellness using a visual analog scale from 0-10 with 0 being extremely low and 10 being extremely high
Self-reported Wellness Assessment | 4 week timepoint
  Subjects report their self-reported wellness using a visual analog scale from 0-10 with 0 being extremely low and 10 being extremely high
Blood Pressure | baseline
  Blood pressure (diastolic and systolic) is measured using an automated machine
Blood Pressure | 4 week timepoint
  Blood pressure (diastolic and systolic) is measured using an automated machine
Heart Rate | baseline
  Heart Rate is measured using an automated machine
Heart Rate | 4 week timepoint
  Heart Rate is measured using an automated machine

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States